CLINICAL TRIAL: NCT02683720
Title: Evaluating the Efficacy of a Novel Oral Supplement in Tackling Malnutrition in the Elderly
Acronym: ProMO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wageningen University (Other)
Collaborators: Vitalnext (Unknown)
Responsible Party: Principal Investigator, Lisette de Groot, MSc PhD Prof, Wageningen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NL56873.081.16
Record Dates: First submitted 2016-02-12; First posted 2016-02-17 (Estimated); Last update posted 2016-07-21 (Estimated); Status verified 2016-07

CONDITIONS: Malnutrition; Muscle Health
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ONS1 (Experimental): new product
  Interventions: Dietary Supplement: ONS
- ONS2 (Active Comparator): usual care
  Interventions: Dietary Supplement: ONS

INTERVENTIONS:
Dietary Supplement: ONS — randomized clinical trial involving different ONS strategies

SUMMARY:
ProMO aims to investigate the effectiveness of a newly developed ONS in increasing body weight, muscle mass and function in malnourished elderly compared to standard care.

ELIGIBILITY:
Inclusion Criteria:

* age 65+
* at risk of malnutrition/ malnourished

Exclusion Criteria:

* • Mental status that is incompatible with the proper conduct of the study

  * Illness of such severity that life expectancy is considered to be less than 12 months
  * Use of diabetes medication (e.g. insulin, methformin)
  * Use of an oral nutritional supplement in the previous three months
  * Participating in any regular exercise training program (≥2h/w)
  * Renal insufficiency (eGFR <30 mL/min/1.73 m2)
  * Unstable organ failure or organ failure necessitating a special diet
  * Chronic corticosteroids use
  * Recent (previous 2 months) use of antibiotics
  * Recent (previous 3 months) change in habitual medication use (e.g statins and thyroxin)
  * Recent blood donation (<1 month prior to Day 01 of the study)
  * Not willing or afraid to give blood during the study
  * Allergic or sensitive for milk proteins
  * Reported vegan or macrobiotic life-style
  * Drug and/or alcohol abuse (current consumption of more than 21 alcoholic drinks per week)
  * Individual unable to give informed consent
  * Current participation in other research from the Division of Human Nutrition
  * Not having a general practitioner
  * Personnel of Wageningen University, department of Human Nutrition, their partner and their first and second degree relatives

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 82 (Estimated)
Dates: Start 2016-07; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
lean body mass | 12 weeks

SECONDARY OUTCOMES:
body weight | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Wageningen University, Wageningen, Netherlands

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Grootswagers P, Smeets E, Oteng AB, Groot L. A novel oral nutritional supplement improves gait speed and mitochondrial functioning compared to standard care in older adults with (or at risk of) undernutrition: results from a randomized controlled trial. Aging (Albany NY). 2021 Apr 2;13(7):9398-9418. doi: 10.18632/aging.202912. Epub 2021 Apr 2. PMID 33799307